CLINICAL TRIAL: NCT06161233
Title: Pilot Study of the eHealth Application "Cancer Patients Better Life Experience" (CAPABLE) - Italy
Acronym: CAPABLE-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: University of Pavia (Other); Policlinico di Bari Ospedale Giovanni Paolo XXIII (Unknown); Biomeris srl (Unknown); The Netherlands Cancer Institute NKI (Unknown); University of Haifa (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); IBM Research (Unknown); Bitsens JSC (Unknown); Poznań University of Technology (Unknown); Deontics LTD (Unknown); Associazione Italiana Malati di Cancro AIMAC (Unknown); Universidad Politecnica de Madrid (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CAPABLE-IT
Record Dates: First submitted 2023-11-30; First posted 2023-12-07 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Renal Cell Carcinoma Metastatic; Breast Cancer; Head and Neck Cancer; Thyroid Cancer; Ovary Cancer; Lung Cancer; Stomach Cancer
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms; Thyroid Neoplasms; Ovarian Neoplasms; Lung Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAPABLE cohort (Experimental): Group that receives the CAPABLE mobile application and a smartwatch during treatment
  Interventions: Device: CAPABLE cohort

INTERVENTIONS:
Device: CAPABLE cohort — The CAPABLE cohort receives the mobileapplication and a multi-sensorial smartwatch (ASUS VivoWatch 5 HC-B05). Patients will be asked to use the system for at least 6 months. The CAPABLE app serves three main functionalities for the patient: symptom monitoring, information needs fulfilment and interventions to improve mental- and physical wellbeing

SUMMARY:
The purpose of the CAPABLE study is to compare health-related quality of life in renal cell carcinoma patients who use or do not use a mobile-based application to monitor adverse events for cancer treatment at home. As secondary objectives, the study investigates the usability of the system and its generalizability to other cancer types

DETAILED DESCRIPTION:
The study is designed as a prospectively enrolling, quasi-experimental cohort study in cancer patients, eligible for systemic treatment.

The CAPABLE cohort will receive the smartphone application and a multi-sensorial smartwatch (ASUS VivoWatch 5 HC-B05). Patients will be asked to use the system for at least 6 months after enrollment. If, after 6 months, a patient wants to keep using the system, he will be allowed to do so, until the end of the study. Questionnaires on health-related quality of life will be administered to the patients on baseline (T0) and every three months (T1 and T2). Lost to follow-up data will be included in intention-to-treat analysis. Qualitative and quantitative user experience studies will be done at enrollment, after 3 months and at the end of the follow-up period with the CAPABLE system. Results of this interventional study will be compared with a control cohort consisting of renal cell carcinoma patients, recruited in 2021 with the same inclusion criteria as this study population, but receiving standard care (ICSM CE number 2546, dated 13/04/2021 and amended on 09/02/2022).

ELIGIBILITY:
Inclusion Criteria:

* Adults (age >=18 years)
* Sufficient understanding of the Italian language
* Patients or their caregiver (upon patient's consent) can use a smartphone
* Histologically or cytologically confirmed diagnosis of RCC, lung, breast, thyroid o head and neck cancer
* Candidate to systemic treatment (targeted agents, immune checkpoint inhibitors, or a combination of the two)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 at the start of the treatment.

Exclusion Criteria:

* Recruitment and consent denial
* Not able of understanding and complying with the protocol requirements (including basic technological abilities)
* Given the fact that each subject involved in the clinical study must be able to understand and sign the informed consent presented by the researcher, lack of this capability represents a specific exclusion criterion in the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Change in health-related QoL outcomes in RCC patients | 6 months after the enrollment
  The primary objective of this study is to investigate whether HRQoL of RCC patients eligible for systemic treatment can be improved by a patient-centred mobile coaching- and monitoring system

SECONDARY OUTCOMES:
User experience of the CAPABLE system in RCC patients | 6 months after the enrollment
  This study will gather qualitative and quantitative information to quantify usefulness, easiness, acceptability and feasibility of the end users' solutions. The patient app will be assessed also in terms of perceived impact and support derived from the digital technologies. The health professional web application will be evaluated to understand to what extent this can be integrated and adopted in the clinical practice
User experience of the CAPABLE system in other cancer types patients | 6 months after the enrollment
  To evaluate the generalizability of the system on other cancer types, the user experience study is performed also on patients with cancer types different from RCC (e.g Breast, Ovary, Head&Neck cancer). The patient app will be assessed also in terms of perceived impact and support derived from the digital technologies. The health professional web application will be evaluated to understand to what extent this can be integrated and adopted in the clinical practice

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri Spa SB, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No